CLINICAL TRIAL: NCT01587118
Title: An Open Label Pilot Study of Adjunctive Asenapine for the Treatment of Posttraumatic Stress Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lori Davis, MD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Forest Laboratories (Industry)
Responsible Party: Sponsor-Investigator, Lori Davis, MD, Associate Chief of Staff, Research and Development Service, Tuscaloosa Research & Education Advancement Corporation
Organization: Tuscaloosa Research & Education Advancement Corporation (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00156
Record Dates: First submitted 2012-04-25; First posted 2012-04-27 (Estimated); Results first posted 2016-12-05 (Estimated); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; Posttraumatic Stress Disorder; Asenapine; Adjunctive; antidepressant; neuroleptic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — asenapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- antidepressant plus asenapine (Experimental): adjunctive asenapine
  Interventions: Drug: Adjunctive asenapine

INTERVENTIONS:
Drug: Adjunctive asenapine — participants who are not responding fully to antidepressant therapy for PTSD will receive adjunctive asenapine (flexible dosing beginning with 5 mg sublingual once per day, titrated up to 10 mg twice per day, as tolerated) for a total of 12 weeks.
  Other Names: asenapine; Saphris

SUMMARY:
This is an open-label pilot study of adjunctive asenapine for the treatment of Posttraumatic Stress Disorder (PTSD) in veterans who have not fully remitted to an adequate trial of standard antidepressant treatment.

DETAILED DESCRIPTION:
Consenting Veterans with the diagnosis of PTSD who have not fully remitted to an adequate trial of standard antidepressant treatment (sertraline, citalopram, escitalopram, fluoxetine, venlafaxine, or mirtazapine) are treated with the addition of open-label asenapine for 12-weeks.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent and acceptable proof of identity.
* Male or female subjects ≥19 to 65 years of age of any race or ethnic origin.
* Not currently pregnant, breastfeeding or planning on becoming pregnant; use of contraception as follows:
* Males - those that are sexually active must use a double barrier method of contraception (condom with spermicide) from the first dose of asenapine until 12 weeks after last dose of asenapine
* Women of child-bearing potential - must have a negative urine pregnancy test and confirmed (by the investigator) use of a highly effective form of birth control for 3 months before enrollment and until 12 weeks after their last dose of asenapine.
* Women of non-child bearing potential - women who are either permanently sterilized (hysterectomy, bilateral oophorectomy and bilateral salpingectomy but excluding bilateral tubal occlusion) or who are postmenopausal.
* Diagnosis of PTSD (DSM-IV-TR criteria; confirmed by MINI and CAPS).
* Total CAPS score > 45.
* Currently taking an approved antidepressant at acceptable dose for 8 weeks or more with non-remission of symptoms.
* No substance use disorders of dependence (except for nicotine, caffeine) in previous 4 wks.
* No substance use disorders of abuse (except for nicotine and caffeine) in the previous 2 wks.
* Physical and laboratory panel (within past one year) are within normal limits or not clinically significant

Exclusion Criteria:

* Lifetime history of bipolar I, schizophrenia, schizoaffective or cognitive disorders (assessed by the MINI)
* Actively considering plans of suicide or homicide (assessed by clinical interview)
* Psychotic symptoms that in the investigator's opinion impair the subject's ability to give informed consent
* A contraindication to the use of asenapine or antidepessant
* Intolerable side effects or allergic reaction to asenapine or the current antidepressant
* Women planning to become pregnant or breastfeed during the study
* Clinically significant unstable or severe medical condition that would contraindicate study participation or expose them to an undue risk of a significant adverse event, including but not limited to: unstable or severe hepatic, renal, respiratory, cardiovascular, endocrine, neurologic, or hematologic disease; hypo- or hyperthyroidism, unless the condition has been stabilized; or a history of seizures (except for a single childhood febrile seizure, posttraumatic, or alcohol withdrawal). The following are exclusionary: platelets < 75,000/mm; hemoglobin <9g/dL; neutrophils, absolute < 1000/mm; LFTs > 3x upper limit; creatinine > 2 mg/dL; diastolic BP < 60 or > 110mmHg; EKG QTc > 475 msec.
* In regard to vulnerable patient populations, persons with dementia, minors (<age 19), the elderly (>age 65), prisoners and the terminally ill are excluded.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori L Davis, MD, Principal Investigator — Tuscaloosa Research & Education Advancement Corporation
Locations (1):
- Tuscaloosa VA Medical Center, Tuscaloosa, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
No sharing of individual participant data

REFERENCES:
- [Result] Pilkinton P, Berry C, Norrholm S, Bartolucci A, Birur B, Davis LL. An Open Label Pilot Study of Adjunctive Asenapine for the Treatment of Posttraumatic Stress Disorder. Psychopharmacol Bull. 2016 Aug 15;46(2):8-17. doi: 10.64719/pb.4349. PMID 27738377

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Antidepressant Plus Asenapine
Started | 18 (31 signed consent and 18 were deemed eligible and initiated treatment with adjunctive asenapine.)
Completed | 11
Not Completed | 7
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 2
Not completed — Relocation | 1
Not completed — nonresponse | 1

BASELINE CHARACTERISTICS:
Arm/Group | Antidepressant Plus Asenapine
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 6
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Clinical Administered PTSD Scale (CAPS) Total
Description: CAPS is the clinician rating of posttraumatic stress disorder (PTSD) symptoms; higher scores indicate higher severity of PTSD; 17-item score range 0 to 136. Blake DD, Weathers FW, Nagy LM, et al. The development of a Clinician-Administered PTSD Scale. J Trauma Stress 1995; 8:75-90.
Time Frame: baseline, week 4, 8, and 12
Population: Open label treatment, all participants included.Overall change in values from baseline to week 12, including weeks 4 and 8, using a simple one-way analysis of variance; because the sample size was small, p-values for the paired t-test and one-way results were recalculated using the signed rank test and Kruskal Wallis procedure, respectively
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Antidepressant Plus Asenapine
Number analyzed (Participants) | 18
units on a scale | -39 (18.4)
Statistical Analysis 1: Comparison: Antidepressant Plus Asenapine; Test type: Superiority or Other; p < .0001, ANOVA — The a priori threshold for statistical significance was p</= 0.05; Change from baseline analyses were conducted using simple one-way analysis of variance; and were recalculated using the Kruskal Wallis procedure

2. Secondary Outcome: Change From Baseline in Brief Psychiatric Rating Scale (BPRS)
Description: BPRS is the clinician rating of psychiatric symptoms; higher score indicates higher severity; 18-items scored 1-7; highest score 126. Overall JE and Gorham DR. The Brief Psychiatric Rating Scale (BPRS): recent developments in ascertainment and scaling. Psychopharmacol Bulletin 1993; 24:97-99.
Time Frame: Baseline, week 4, 8, 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Antidepressant Plus Asenapine
Number analyzed (Participants) | 18
units on a scale | -15.5 (9.3)
Statistical Analysis 1: Comparison: Antidepressant Plus Asenapine; Test type: Superiority or Other; p = .0006, ANOVA — The a priori threshold for statistical significance was p</= 0.05; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the 12 weeks of active study participation; Serious adverse events were collected for the 12 weeks of study and one additional post-study month.
Arm/Group | Antidepressant Plus Asenapine
Serious Adverse Events (participants affected / at risk) | 1/18
Other Adverse Events (participants affected / at risk) | 6/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antidepressant Plus Asenapine (N=18)
Psychiatric hospitalization (Psychiatric disorders) | 1 (1) — One participant was hospitalized on psychiatric unit in the month following study exit while not on asenapine; Unrelated SAE.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antidepressant Plus Asenapine (N=18)
sedation with syncope (Nervous system disorders) | 1 (1) — sedation with syncope day 1 while on asenapine 5mg/d; stopped study medication.
weight gain (Metabolism and nutrition disorders) | 1 (1) — weight gain at week 4 on 5mg/d asenapine; stopped asenapine
sedation (Nervous system disorders) | 2 (2) — sedation at week 4 in one participant and sedation at week 12 in one participant; both stopped asenapine.
extrapyramidal side effect (Nervous system disorders) | 1 (1) — extrapyramidal side effects at week 12 on 20mg/d asenapine; stopped asenapine
Headache (Nervous system disorders) | 1 (1) — On 10mg/d asenapine
sinus infection (Infections and infestations) | 1 (1) — Unrelated to asenapine
upset stomach (Gastrointestinal disorders) | 1 (1) — asenapine 10mg/d
fatigue (General disorders) | 1 (1) — 10mg/d asenapine
agitation (General disorders) | 1 (1) — day 4 on 5mg/d asenapine, stopped asenapine

LIMITATIONS AND CAVEATS:
This study was limited by both the small number of subjects enrolled and its open-label design.

Average dose of asenapine was 13.6 ± 6.4 mg/d; at 12-weeks 15.9 ± 4.9 mg/d.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No